CLINICAL TRIAL: NCT02923921
Title: Randomized Study of AM0010 in Combination With FOLFOX Compared to FOLFOX Alone as Second-line Tx in Pts With Metastatic Pancreatic Cancer That Has Progressed During or Following a First-Line Gemcitabine Containing Regimen
Brief Title: Study of Pegilodecakin (LY3500518) With FOLFOX Compared to FOLFOX Alone Second-line Tx in Participants With Metastatic Pancreatic Cancer
Acronym: Sequoia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ARMO BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17158; J1L-AM-JZGB (Other: Eli Lilly and Company); AM0010-301 (Other: ARMO BioSciences); 2016-003858-33 (EudraCT Number)
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-04-15

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pegilodecakin; AM0010; Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegilodecakin + FOLFOX (Experimental): Pegilodecakin 5 microgram per kilogram (μg/kg) dosed as one of the following 2 fixed doses: 0.4 milligram (mg) for participants weighing ≤80 kg or 0.8 mg for participants weighing>80 kg on Days 1-5 and Days 8-12 subcutaneously (SC) plus FOLFOX [dl-Leucovorin (dl-LV) 400 milligram per meter square (mg/m2) and oxaliplatin 85 mg/m2 followed by bolus 5-fluorouracil (5-FU) 400 mg/m2 and a 46 to 48 hour infusion of 5- FU 2400 mg/m2] initiated on Day 1 of a 14-day cycles for up to 12 cycles or until disease progression. After discontinuation of FOLFOX in the absence of tumor progression [that is (i.e., completion of the planned 12 cycles or unacceptable FOLFOX related toxicity], Pegilodecakin 10µg/kg maintenance treatment administered as one of the 2 fixed doses, either 0.8 mg for participants weighing ≤80 kg or 1.6 mg for participants weighing>80 kg.
  Interventions: Biological: Pegilodecakin; Drug: FOLFOX
- FOLFOX (Active Comparator): FOLFOX (dl-LV 400 mg/m2 and oxaliplatin 85 mg/m2 followed by bolus 5-FU 400 mg/m2 and a 46-hour infusion of 5-FU 2400 mg/m2) initiated on Day 1 of a 14-day cycles for up to 12 cycles or until disease progression.
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Biological: Pegilodecakin — Pegilodecakin plus FOLFOX
  Other Names: LY3500518; AM0010
  Arms: Pegilodecakin + FOLFOX
Drug: FOLFOX — FOLFOX Alone
  Other Names: oxaliplatin; 5-FU; leucovorin

SUMMARY:
To compare the efficacy of pegilodecakin in combination with FOLFOX versus FOLFOX alone in participants with metastatic pancreatic cancer as measured by overall survival.

DETAILED DESCRIPTION:
This is an open-label, multi-center, randomized, Phase 3 study designed to compare the efficacy and safety of pegilodecakin in combination with FOLFOX versus FOLFOX alone in participants with metastatic adenocarcinoma of the pancreas who have progressed on one prior gemcitabine containing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of metastatic pancreatic adenocarcinoma
2. Measurable disease per RECIST v.1.1
3. Participant must have documented tumor progression during or following a gemcitabine containing regimen to treat metastatic disease as established by CT or MRI scan
4. Eastern Cooperative Oncology Group Performance Status of 0 - 1
5. Participant must have completed prior chemotherapy at least 2 weeks (washout period) prior to randomization and recovered from toxicity to Grade 1 or baseline
6. Participants must not have received previous radiation therapy or investigational therapy for the treatment of advanced metastatic disease.
7. Participants having received cytotoxic doses of gemcitabine or any other chemotherapy in the adjuvant setting are not eligible for this study
8. No peripheral neuropathy
9. No known history of dihydropyrimidine dehydrogenase deficiency

Exclusion Criteria:

1. Diagnosis of pancreatic islet neoplasm, acinar cell carcinoma, non- adenocarcinoma (i.e., lymphoma, sarcoma), adenocarcinoma originating from the biliary tree, or cystadenocarcinoma
2. Participant on Coumadin and not willing to change to LMWH or oral Factor II or Xa inhibitor with half-life of less than 24 hours.
3. Participant has received prior treatment with pegilodecakin or fluoropyrimidine/platinum containing regimen
4. Participants who were intolerant of a gemcitabine containing regimen.
5. History of positivity for human immunodeficiency virus
6. Chronic active or active viral hepatitis A, B, or C infection
7. Clinically significant bleeding within two weeks prior to randomization (e.g., gastrointestinal (GI) bleeding, intracranial hemorrhage)
8. Pregnant or lactating women
9. Participants with a history of immune-mediated neurological disorders such as multiple sclerosis, Guillain-Barré or inflammatory CNS/PNS disorders
10. Clinically significant ascites defined as requiring ≥ 1 paracentesis every 2- weeks
11. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e., larger than what is required for placement of central venous access, percutaneous feeding tube, or biopsy),within 28 days prior to randomization or anticipated surgery during the study period
12. Prior history of receiving immune modulators including, but not limited to, anti-CTLA4, anti-PD1, anti-PD-L1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (130):
- United States (57):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cancer Treatment Centers of America, Goodyear, Arizona
  - University of Arizona Cancer Center, Phoenix, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - USC Norris Cancer Hospital, Los Angeles, California
  - TRIO - Translational Research in Oncology-US, Inc., Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Cancer Care Associates Medical Group, Redondo Beach, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Lynn Cancer Institute Ctr for Hem-Onc, Boca Raton, Florida
  - Memorial Regional Hospital/Joe Dimaggio Childrens Hospital, Hollywood, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Watson Clinic, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - UF Health Cancer Center- Orlando Health, Orlando, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Saint Alphonsus Regional Medical Center, Caldwell, Idaho
  - Decatur Memorial Hospital, Decatur, Illinois
  - Fort Wayne Oncology & Hematology, Fort Wayne, Indiana
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - New England Cancer Specialists - Scarborough, Scarborough, Maine
  - Committee on Clinical Investigations (CCI)- Beth Isreal Deaconess Medical Center IRB, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - St Louis Cancer Care, Bridgeton, Missouri
  - Summit Medical Group, Summit, New Jersey
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Winthrop University Hospital, Mineola, New York
  - Duke University Medical Center, Durham, North Carolina
  - Novant Health, Oncology Research Institute, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - US Oncology, The Woodlands, Texas
  - Hope Cancer Center of East Texas, Tyler, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology-Wichital Falls Texoma Cancer Center, Wichita Falls, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - Medical Oncology Associates, PS, Spokane, Washington
  - MultiCare Regional Cancer Center - Auburn, Tacoma, Washington
  - Aurora West Allis Medical Center, Green Bay, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - St Vincent's Hospital, Sydney, New South Wales
  - Warringal Private Hospital, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - St John of God Murdoch Hospital, Murdoch, Western Australia
- Austria (3):
  - Universitätsklinikum Graz, Graz, Styria
  - KH der Barmherzigen Schwestern Linz BetriebsGesmbH, Linz, Upper Austria
  - Universitätsklinikum Salzburg, Salzburg
- Belgium (10):
  - Imeldaziekenhuis, Bonheiden
  - Hospital Universitaire Erasme Brussel, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Grand Hopital de Charleroi-Site Notre-Dame, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge, Kortrijk
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Clinique St Elisabeth Namur, Namur
  - CHU Dinant Godinne - UCL Namur, Yvoir
- Canada (2):
  - Toronto Sunnybrook Regional Cancer Center, Toronto, Ontario
  - McGill University, Montreal, Quebec
- France (4):
  - CHU de Besancon Hopital Jean Minjoz, Besançon
  - Hopital de la Pitie Salpetriere, Paris
  - CHU la Miletrie, Poitiers
  - Hôpital Nord Franche-Comté, Trévenans
- Germany (7):
  - Städtisches Klinikum München, München, Bavaria
  - Kliniken Essen-Mitte Ev. Huyssens-Stiftung, Essen, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Charité Universitätsmedizin Berlin, Berlin
  - St Josef-Hospital Bochum, Bochum
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Klinik Altona, Hamburg
- Italy (11):
  - Istituto Scientifico Romagnolo - Studio e la Cura dei Tumori, Meldola, Forli
  - Fondazione Piemonte l'Oncologia-Istituto Ricerca Cura Cancro, Candiolo, Torino
  - Ospedale le Torrette, Ancona
  - Azienda Ospedaliera Universitaria Ospedale San Martino di Genova, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale Niguarda Ca Granda, Milan
  - AOU dell'Università degli Studi della Campania Luigi Vanvitelli, Naples
  - Istituto Oncologico Veneto, Padua
  - Policlinico San Matteo, Pavia
  - Arcispedale Santa Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Universita Campus Biomedico, Roma
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szp.Kliniczny Przemienienia Panskiego UM im.K.Marcinkowskieg, Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - Wojewodzki Szpital Zespolony, Torun
- South Korea (6):
  - Dong-A University Medical Center, Busan, Busan Gwang'yeogsi
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Severance Hospital Yonsei University Health System, Seoul, Korea
  - Samsung Medical Center, Seoul, Korea
  - Seoul St. Mary's Hospital, Seoul, Korea
  - Asan Medical Center, Seoul
- Spain (14):
  - Hospital Duran I Reynals, Hospitaled de Llobre, Barcelona
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, La Coruna
  - Hospital General Universitario Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital General Yague, Burgos
  - C.H. Regional Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Regional University Hospital in Malaga, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (3):
  - Tri-Service General Hospital, Neihu Taipei
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Hammersmith Hospital, Acton, London
  - Velindre Hospital, Cardiff, South Glamorgan
  - University College London Hospital Foundation Trust, London, Surrey
  - Guys/St. Thomas Hospital, London, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hecht JR, Lonardi S, Bendell J, Sim HW, Macarulla T, Lopez CD, Van Cutsem E, Munoz Martin AJ, Park JO, Greil R, Wang H, Hozak RR, Gueorguieva I, Lin Y, Rao S, Ryoo BY. Randomized Phase III Study of FOLFOX Alone or With Pegilodecakin as Second-Line Therapy in Patients With Metastatic Pancreatic Cancer That Progressed After Gemcitabine (SEQUOIA). J Clin Oncol. 2021 Apr 1;39(10):1108-1118. doi: 10.1200/JCO.20.02232. Epub 2021 Feb 8. PMID 33555926

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Participant Flow, participants who completed were those who died due to any cause or were alive and on study at conclusion but off treatment.
Groups:
- Pegilodecakin + FOLFOX: Pegilodecakin 5 microgram per kilogram (μg/kg) dosed as one of the following 2 fixed doses: 0.4 milligram (mg) for participants weighing less than or equal to (≤) 80 kg or 0.8 mg for participants weighing greater than (>) 80 kg on Days 1-5 and Days 8-12 subcutaneously (SC) plus FOLFOX [dl-Leucovorin (dl-LV) 400 milligram per meter square (mg/m2) and oxaliplatin 85 mg/m2 followed by bolus 5-fluorouracil (5-FU) 400 mg/m2 and a 46 to 48 hour infusion of 5- FU 2400 mg/m2] initiated on Day 1 of a 14-day cycles for up to 12 cycles or until disease progression. After discontinuation of FOLFOX in the absence of tumor progression [that is (i.e., completion of the planned 12 cycles or unacceptable FOLFOX related toxicity], Pegilodecakin 10µg/kg maintenance treatment administered as one of the 2 fixed doses, either 0.8 mg for participants weighing ≤80 kg or 1.6 mg for participants weighing>80 kg.
- FOLFOX: FOLFOX (dl-LV 400 mg/m2 and oxaliplatin 85 mg/m2 followed by bolus 5- FU 400 mg/m2 and a 46-hour infusion of 5-FU 2400 mg/m2) initiated on Day 1 of a 14-day cycles for up to 12 cycles or until disease progression.
Period: Overall Study
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX
Started | 283 | 284
Received at Least 1 Dose of Study Drug | 278 | 251
Safety Population | 278 | 251
Completed | 230 | 227
Not Completed | 53 | 57
Not completed — Sponsor Decision | 39 | 38
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Unknown, Not Collected | 7 | 6

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Pegilodecakin + FOLFOX: Pegilodecakin 5 μg/kg dosed as one of the following 2 fixed doses: 0.4 mg for participants weighing ≤80 kg or 0.8 mg for participants weighing>80 kg on Days 1-5 and Days 8-12 subcutaneously (SC) plus FOLFOX [dl-Leucovorin (dl-LV) 400 mg/m2 and oxaliplatin 85 mg/m2 followed by bolus 5-fluorouracil (5-FU) 400 mg/m2 and a 46 to 48 hour infusion of 5- FU 2400 mg/m2] initiated on Day 1 of a 14-day cycles for up to 12 cycles or until disease progression. After discontinuation of FOLFOX in the absence of tumor progression [that is (i.e., completion of the planned 12 cycles or unacceptable FOLFOX related toxicity], Pegilodecakin 10µg/kg maintenance treatment administered as one of the 2 fixed doses, either 0.8 mg for participants weighing ≤80 kg or 1.6 mg for participants weighing>80 kg.
- Total: Total of all reporting groups
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX | Total
Number analyzed (Participants) | 283 | 284 | 567
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.0) | 64.1 (9.9) | 64.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 132 | 267
  Male | 148 | 152 | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 263 | 265 | 528
  Unknown or Not Reported | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 59 | 55 | 114
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 8 | 16
  White | 207 | 213 | 420
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 93 | 89 | 182
  United Kingdom | 5 | 4 | 9
  Spain | 42 | 31 | 73
  Canada | 2 | 7 | 9
  South Korea | 48 | 41 | 89
  Austria | 3 | 10 | 13
  Belgium | 17 | 19 | 36
  Taiwan | 5 | 10 | 15
  Poland | 8 | 5 | 13
  Italy | 28 | 39 | 67
  France | 9 | 2 | 11
  Australia | 14 | 16 | 30
  Germany | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of randomization to the date of death (due to any cause). For participants whose last known status is alive at the data cutoff date for the analysis, time will be censored as the last contact date prior to the data cutoff date.
Time Frame: Randomization to date of death from any cause (Up To 30 Months)
Population: All randomized participants. The number of participants censored were Pegilodecakin + FOLFOX = 63 and FOLFOX = 73.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX
Number analyzed (Participants) | 283 | 284
Months | 5.78 [5.45 to 6.64] | 6.28 [5.62 to 7.39]
Statistical Analysis 1: Comparison: Pegilodecakin + FOLFOX vs FOLFOX; The primary test to compare overall survival between treatment arms was the two-sided log-rank test, stratified by region and prior therapy. The estimate of the hazard ration (HR) - (Pegilodecakin + FOLFOX Arm / FOLFOX Arm) and the corresponding 95% CI was computed using a Cox proportional hazards model stratified by randomization stratification factors. Randomization stratification factors were based on the data recorded in interactive voice response system (IVRS); Test type: Superiority; p = 0.6565, Log Rank; Hazard Ratio (HR) = 1.045, 95% CI 2-sided [0.863 to 1.265]

2. Secondary Outcome: Progression Free Survival
Description: PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant did not have a complete baseline disease assessment, then PFS was censored at the enrollment date, regardless whether or not objectively determined PD or death had been observed for the participant.
Time Frame: Randomization to Progressive Disease (PD) or Date of Death (Up To 30 Months)
Population: All randomized participants. The number of participants censored were Pegilodecakin + FOLFOX = 45 and FOLFOX = 86.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX
Number analyzed (Participants) | 283 | 284
Months | 2.14 [1.94 to 3.38] | 2.10 [1.94 to 3.25]
Statistical Analysis 1: Comparison: Pegilodecakin + FOLFOX vs FOLFOX; The estimate of hazard ratio (HR) was stratified by region and prior therapy; Test type: Superiority; p = 0.8144, Log Rank; Hazard Ratio (HR) = 0.981, 95% CI 2-sided [0.808 to 1.190]

3. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)] That Assessed by Investigator
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. Participants who discontinued study treatment (for reasons other than progression) before entering concurrent phase were considered to have non-evaluable response.
Time Frame: Randomization to PD (Up To 30 Months)
Population: All randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX
Number analyzed (Participants) | 283 | 284
Percentage of participants | 4.6 | 5.6
Statistical Analysis 1: Comparison: Pegilodecakin + FOLFOX vs FOLFOX; Test type: Superiority; p = 0.7044, Cochran-Mantel-Haenszel — P-value is calculated by Exact Cochran-Mantel-Haenszel test stratified by the randomization strata Prior Therapy - interactive voice response system (IVRS), Geographic Region - IVRS; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.7]

4. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD): Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization to Objective Progressive Disease or Start of New Anti-Cancer Therapy (Up To 30 Months)
Population: All randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX
Number analyzed (Participants) | 283 | 284
Percentage of participants | 42.8 | 36.6
Statistical Analysis 1: Comparison: Pegilodecakin + FOLFOX vs FOLFOX; Test type: Superiority; p = 0.1463, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.9 to 1.8]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization to Progressive Disease (PD) or Date of Death (Up To 30 Months)
Population: All randomized participants who achieved an objective response of CR or PR. The number of participants censored were Pegilodecakin + FOLFOX = 4 and FOLFOX = 7.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX
Number analyzed (Participants) | 13 | 16
Months | 4.99 [3.45 to 7.06] | 5.17 [3.75 to 5.72]
Statistical Analysis 1: Comparison: Pegilodecakin + FOLFOX vs FOLFOX; The estimate of hazard ratio (HR) was stratified by region and prior therapy; Test type: Superiority; p = 0.9952, Log Rank; Hazard Ratio (HR) = 1.008, 95% CI 2-sided [0.370 to 2.741]

6. Secondary Outcome: Percentage of Participants Alive at 1 Year (12-Month Survival Rate)
Description: The 12-month survival rate is defined as the percentage of participants who have not died 12 months after the date of randomization.
Time Frame: From randomization to until the date of first documented date of death from any cause within 12 months
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX
Number analyzed (Participants) | 283 | 284
Percentage of participants | 14.7 [10.2 to 19.9] | 19.1 [14.1 to 24.7]
Statistical Analysis 1: Comparison: Pegilodecakin + FOLFOX vs FOLFOX; Test type: Superiority; p = 0.2298, Log Rank; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-11.6 to 2.8]

ADVERSE EVENTS:
Time Frame: Baseline Up To 36 Months
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Pegilodecakin + FOLFOX | FOLFOX
All-Cause Mortality (participants affected / at risk) | 217/278 | 188/251
Serious Adverse Events (participants affected / at risk) | 123/278 | 95/251
Other Adverse Events (participants affected / at risk) | 271/278 | 240/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pegilodecakin + FOLFOX (N=278) | FOLFOX (N=251)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 11 (14) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 5 (5)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8) | 5 (5)
Asthenia (General disorders) | 2 (2) | 1 (1)
Euthanasia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 2 (2)
General physical health deterioration (General disorders) | 3 (3) | 2 (3)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 13 (15) | 7 (7)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 6 (8) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 2 (3) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3) | 3 (3)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 2 (2)
Biliary tract infection (Infections and infestations) | 3 (3) | 1 (4)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Cholangitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 4 (5) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (8) | 4 (4)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 10 (10) | 4 (4)
Septic shock (Infections and infestations) | 4 (7) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 4 (6)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 2 (3) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Device failure (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 3 (3) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1/144 (1) | 0/134 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic embolus (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 2 (2)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegilodecakin + FOLFOX (N=278) | FOLFOX (N=251)
Anaemia (Blood and lymphatic system disorders) | 107 (204) | 38 (56)
Neutropenia (Blood and lymphatic system disorders) | 58 (118) | 41 (65)
Thrombocytopenia (Blood and lymphatic system disorders) | 99 (296) | 28 (42)
Abdominal distension (Gastrointestinal disorders) | 18 (22) | 14 (15)
Abdominal pain (Gastrointestinal disorders) | 82 (114) | 58 (82)
Abdominal pain upper (Gastrointestinal disorders) | 20 (34) | 14 (17)
Ascites (Gastrointestinal disorders) | 28 (35) | 19 (20)
Constipation (Gastrointestinal disorders) | 79 (93) | 59 (70)
Diarrhoea (Gastrointestinal disorders) | 70 (104) | 71 (101)
Dyspepsia (Gastrointestinal disorders) | 21 (23) | 14 (16)
Flatulence (Gastrointestinal disorders) | 14 (15) | 4 (6)
Nausea (Gastrointestinal disorders) | 126 (217) | 106 (160)
Stomatitis (Gastrointestinal disorders) | 27 (37) | 40 (48)
Vomiting (Gastrointestinal disorders) | 80 (122) | 69 (106)
Asthenia (General disorders) | 76 (151) | 45 (105)
Fatigue (General disorders) | 105 (181) | 74 (108)
Injection site erythema (General disorders) | 18 (18) | 0 (0)
Oedema peripheral (General disorders) | 41 (49) | 22 (25)
Pyrexia (General disorders) | 56 (82) | 36 (51)
Aspartate aminotransferase increased (Investigations) | 12 (17) | 14 (22)
Blood alkaline phosphatase increased (Investigations) | 21 (28) | 15 (20)
Blood bilirubin increased (Investigations) | 19 (28) | 10 (12)
Neutrophil count decreased (Investigations) | 47 (84) | 30 (51)
Platelet count decreased (Investigations) | 59 (163) | 26 (51)
Weight decreased (Investigations) | 14 (17) | 25 (34)
Decreased appetite (Metabolism and nutrition disorders) | 97 (132) | 77 (100)
Dehydration (Metabolism and nutrition disorders) | 12 (22) | 14 (19)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (20) | 10 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 (28) | 10 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (37) | 29 (39)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (15) | 16 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 37 (44) | 32 (39)
Dizziness (Nervous system disorders) | 19 (23) | 8 (9)
Dysgeusia (Nervous system disorders) | 19 (22) | 9 (11)
Headache (Nervous system disorders) | 18 (24) | 17 (20)
Neuropathy peripheral (Nervous system disorders) | 40 (50) | 38 (62)
Neurotoxicity (Nervous system disorders) | 13 (25) | 15 (30)
Paraesthesia (Nervous system disorders) | 24 (34) | 17 (44)
Peripheral sensory neuropathy (Nervous system disorders) | 31 (48) | 29 (35)
Polyneuropathy (Nervous system disorders) | 9 (13) | 14 (25)
Insomnia (Psychiatric disorders) | 14 (14) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 19 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (41) | 15 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (24) | 8 (11)
Rash (Skin and subcutaneous tissue disorders) | 23 (34) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT02923921/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT02923921/SAP_001.pdf